CLINICAL TRIAL: NCT04436510
Title: HEALEY ALS Platform Trial - Regimen B Verdiperstat
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merit E. Cudkowicz, MD (Other)
Collaborators: Biohaven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Merit E. Cudkowicz, MD, Chief, Neurology Department, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P003518B
Record Dates: First submitted 2020-06-01; First posted 2020-06-18 (Actual); Results first posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Placebo-Controlled; Double-Blind; Regimen Specific Appendix; Lou Gehrig's Disease; Verdiperstat; Biohaven Pharmaceuticals
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Verdiperstat (Experimental): Verdiperstat is administered twice daily p.o. for 24 weeks.
  Interventions: Drug: Verdiperstat
- Matching Placebo (Placebo Comparator): Matching placebo is administered twice daily p.o. for 24 weeks.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Matching Placebo — Drug: Matching Placebo
  Administration: Oral
  Dose: two tablets twice daily
  Arms: Matching Placebo
Drug: Verdiperstat — Drug: Verdiperstat
  Administration: Oral
  Dose: 600mg twice daily
  Arms: Verdiperstat

SUMMARY:
The HEALEY ALS Platform Trial is a perpetual multi-center, multi-regimen clinical trial evaluating the safety and efficacy of investigational products for the treatment of ALS.

Regimen B will evaluate the safety and efficacy of a single study drug, verdiperstat, in participants with ALS.

DETAILED DESCRIPTION:
The HEALEY ALS Platform Trial is a perpetual multi-center, multi-regimen clinical trial evaluating the safety and efficacy of investigational products for the treatment of ALS. This trial is designed as a perpetual platform trial. This means that there is a single Master Protocol dictating the conduct of the trial. The HEALEY ALS Platform Trial Master Protocol is registered as NCT04297683.

Once a participant enrolls into the Master Protocol and meets all eligibility criteria, the participant will be eligible to be randomized into any currently enrolling regimen. All participants will have an equal chance of being randomized to any currently enrolling regimen.

If a participant is randomized to Regimen B - Verdiperstat, the participant will complete a screening visit to assess additional Regimen B eligibility criteria. Once Regimen B eligibility criteria are confirmed, participants will complete a baseline assessment and be randomized in a 3:1 ratio to either active Verdiperstat or matching placebo.

Regimen B will enroll by invitation as participants may not choose to enroll in Regimen B. Participants must first enroll into the Master Protocol and be eligible to participate in the Master Protocol before being able to be randomly assigned to Regimen B.

For a list of enrolling sites, please see the HEALEY ALS Platform Trial Master Protocol under NCT04297683.

ELIGIBILITY:
Inclusion Criteria:

* No additional inclusion criteria beyond the inclusion criteria specified in the Master Protocol (NCT NCT04297683).

Exclusion Criteria:

* The following exclusion criteria are in addition to the exclusion criteria specified in the Master Protocol (NCT NCT04297683).

  1. Participants who are taking strong inhibitors of CYP1A2 (i.e., ciprofloxacin, enoxacin, fluvoxamine, zafirlukast) for chronic/long-term use defined as more than two weeks.
  2. Participants who are taking strong inhibitors of CYP3A4 (i.e., conivaptan, itraconazole, ketoconazole, posaconazole, troleandomycin, voriconazole, clarithromycin, diltiazem, idelalisib, nefazodone, and certain antiviral agents [cobicistat, danoprevir, ritonavir, elvitegravir, indinavir, lopinavir, paritaprevir, ombitasavir, dasabuvir, saquinavir, tipranavir, nelfinavir]) for chronic/long-term use defined as more than two weeks. Note: Topical antifungal use is not exclusionary. Participants should not consume large quantities of grapefruit juice (more than 8oz per day) on a regular basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merit Cudkowicz, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Healey Center for ALS at Mass General, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Writing Committee for the HEALEY ALS Platform Trial; Andrews J, Paganoni S, Macklin EA, Chibnik LB, Quintana M, Saville BR, Detry MA, Vestrucci M, Marion J, McGlothlin A, Young E, Chase M, Pothier L, Harkey B, Yu H, Sherman A, Shefner J, Hall M, Kittle G, Connolly MR, Berry JD, D'Agostino D, Tustison E, Giacomelli E, Scirocco E, Alameda G, Locatelli E, Ho D, Quick A, Heitzman D, Ajroud-Driss S, Appel SH, Shroff S, Katz J, Felice K, Maragakis NJ, Simmons Z, Goutman SA, Olney N, Miller T, Fernandes JA, Ilieva H, Jawdat O, Weiss MD, Foster L, Vu T, Ladha S, Owegi MA, Newman DS, Arcila-Londono X, Jackson CE, Swenson A, Heiman-Patterson T, Caress J, Fee D, Peltier A, Lewis R, Rosenfeld J, Walk D, Johnson K, Elliott M, Kasarskis EJ, Rutkove S, McIlduff CE, Bedlack R, Elman L, Goyal NA, Rezania K, Twydell P, Benatar M, Glass J, Cohen JA, Jones V, Zilliox L, Wymer JP, Beydoun SR, Shah J, Pattee GL, Martinez-Thompson J, Nayar S, Granit V, Donohue M, Grossman K, Campbell DJ, Qureshi IA, Cudkowicz ME, Babu S. Verdiperstat in Amyotrophic Lateral Sclerosis: Results From the Randomized HEALEY ALS Platform Trial. JAMA Neurol. 2025 Apr;82(4):333-343. doi: 10.1001/jamaneurol.2024.5249. Epub 2025 Feb 17. PMID 40067754

RESULTS

PARTICIPANT FLOW:
Groups:
- Verdiperstat: Verdiperstat is administered twice daily p.o. for 24 weeks.
  Verdiperstat: Drug: Verdiperstat
  Administration: Oral
  Dose: 600mg twice daily
- Matching Placebo: Matching placebo is administered twice daily p.o. for 24 weeks.
  Matching Placebo: Drug: Matching Placebo
  Administration: Oral
  Dose: two tablets twice daily
Period: Overall Study
Arm/Group | Verdiperstat | Matching Placebo
Started | 126 | 41
Completed | 95 | 35
Not Completed | 31 | 6

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population includes only placebo participants from the Regimen B Efficacy Regimen Only (ERO) sample; shared placebo participants from other regimens are not included in the Baseline Analysis Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Verdiperstat | Matching Placebo | Total
Number analyzed (Participants) | 126 | 41 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (11.54) | 57.3 (11.07) | 57.9 (11.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 12 | 59
  Male | 79 | 29 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 0 | 8
  Not Hispanic or Latino | 116 | 41 | 157
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 116 | 37 | 153
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
El Escorial Diagnosis [Count of Participants; unit: Participants]
  Clinically Definite ALS | 45 | 18 | 63
  Clinically Probable ALS | 53 | 11 | 64
  Clinically Probable ALS - Laboratory Supported | 20 | 8 | 28
  Clinically Possible ALS | 8 | 4 | 12
Time Since Symptom onset at Baseline [Mean (Standard Deviation); unit: months] | 21.2 (8.93) | 22.5 (7.91) | 21.5 (8.69)
Delay in ALS Symptom Onset and Diagnosis [Mean (Standard Deviation); unit: months] | 10.5 (5.96) | 10.5 (6.15) | 10.5 (5.99)
ALS Onset Location [Count of Participants; unit: Participants]
  Axial | 1 | 2 | 3
  Bulbar | 20 | 7 | 27
  Generalized | 1 | 0 | 1
  Limb | 103 | 32 | 135
  Respiratory | 1 | 0 | 1
Baseline Edaravone Use [Count of Participants; unit: Participants]
  Yes | 28 | 11 | 39
  No | 98 | 30 | 128
Baseline Riluzole Use [Count of Participants; unit: Participants]
  Yes | 95 | 31 | 126
  No | 31 | 10 | 41
ALSFRS-R Total Score [Mean (Standard Deviation); unit: scores on a scale] — The ALS Functional Rating Scare-Revised (ALSFRS-R) measures 12 aspects of physical function. Each of the 12 questions assessing distinct functional ability is scored from4(normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Patients with higher scores have more physical function.
  scores on a scale | 34.3 (6.45) | 34.3 (6.88) | 34.3 (6.54)
Change in ALSFRS-R prior to Baseline [Mean (Standard Deviation); unit: points per month] — The ALS Functional Rating Scare-Revised (ALSFRS-R) measures 12 aspects of physical function. Each of the 12 questions assessing distinct functional ability is scored from4(normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0.
  Baseline decline in ALSFRS-R was calculated as 48minus the ALSFRS-R total score at Baseline. The difference between 48 and ALSFRS-R total score at Baseline is divided by the number of months between onset of weakness due to ALS and the date of Baseline.
  A higher number indicates greater decline.
  points per month | 0.75 (0.499) | 0.64 (0.303) | 0.72 (0.461)
SVC [Mean (Standard Deviation); unit: Percent Predicted] — Population: Number analyzed in row differs from overall number due to missing data.
  Percent Predicted
    number analyzed (Participants) | 121 | 39 | 160
    (all) | 77.2 (20.37) | 74.5 (17.50) | 76.6 (19.69)
Kings Stage [Count of Participants; unit: Participants] — The King's ALS Clinical Staging System is a 4-level ordinal scale with the first three levels indicating the number (1, 2, or 3) of distinct central nervous system regions (bulbar, upper limb, and lower limb) with neuromuscular dysfunction. Level 4a indicates nutritional failure and level 4b indicates respiratory failure. Higher scores indicate a worse disease state.
  Participants
    1 Region with Neuromuscular Dysfunction | 13 | 9 | 22
    2 Regions with Neuromuscular Dysfunction | 39 | 10 | 49
    3 Regions with Neuromuscular Dysfunction | 36 | 14 | 50
    4a/b Nutritional/Respiratory Failure | 2 | 0 | 2
    4b Respiratory Failure | 36 | 8 | 44
Weight [Mean (Standard Deviation); unit: kg] | 78.7 (17.44) | 82.4 (18.66) | 79.6 (17.76)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.4 (5.13) | 27.1 (4.89) | 26.6 (5.07)
Serum Creatinine Concentration [Mean (Standard Deviation); unit: mg/dL] | 0.7 (0.17) | 0.7 (0.17) | 0.7 (0.17)
Neurofilament Light (NfL) Protein in Serum [Mean (Standard Deviation); unit: ng/L] — Population: Number analyzed in row differs from overall number due to missing data.
  ng/L
    number analyzed (Participants) | 124 | 40 | 164
    (all) | 92.3 (75.27) | 65.8 (25.60) | 85.9 (67.55)

OUTCOME MEASURES:

1. Primary Outcome: Disease Progression as Assessed by the ALSFRS-R-Slope
Description: Change in disease severity as measured by the ALS Functional Rating Scale-Revised (ALSFRS-R) total score using a Bayesian repeated measures model that accounts for loss to follow-up due to mortality. Each of 12 questions assessing distinct functional ability is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Patients with higher scores have more physical function.
Time Frame: Baseline to 24 Weeks
Population: Outcome measure data was analyzed using the Full Analysis Set, which included shared placebo from other regimens, as pre-specified in the Regimen Statistical Analysis Plan. Regimen A Zilucoplan (NCT04436497) and Regimen C CNM-Au8 (NCT04414345) contributed placebo participants into the shared placebo cohort used for analysis.
Measure: Mean (Standard Deviation); unit: ALSFRS-R total score points per month
Arm/Group | Verdiperstat | Matching Placebo
Number analyzed (Participants) | 126 | 122
ALSFRS-R total score points per month | -1.02 (0.091) | -1.05 (0.086)
Statistical Analysis 1: Comparison: Verdiperstat vs Matching Placebo; Test type: Superiority; Bayesian shared-parameter model — Posterior probability that the disease rate ratio (DRR) is less than 1 (i.e. verdiperstat slowed progression) was 0.57467. NOTE: p-value is not provided for Bayesian model; A Bayesian shared-parameter model of change in disease severity as measured by ALSFRS-R total score and mortality; Disease Rate Ratio = 0.98, 95% CI 2-sided [0.769 to 1.237], Standard Deviation 0.118 — DDR <1 imply slowing of disease progression by verdiperstat relative to placebo. Note: reported "Confidence Interval" is actually a Bayesian credible interval; The model includes covariates for baseline use of edaravone, baseline use of riluzole, months since onset of symptoms, and pre-baseline slope of ALSFRS-R, and random effects for regimen and participant-specific slopes

2. Primary Outcome: Mortality Even Rate
Description: Mortality is defined as death or death equivalent. A participant is determined to meet the criteria of death equivalent if permanent assisted ventilation (PAV) is used for more than 22 hours per day for more than seven days in a row. The rate of mortality was estimated from a Bayesian shared-parametric model that assumed exponentially distributed survival times.
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events per month
Arm/Group | Verdiperstat | Matching Placebo
Number analyzed (Participants) | 126 | 122
events per month | 0.011 (0.003) | 0.012 (0.003)

3. Secondary Outcome: Respiratory Function
Description: Change in respiratory function over time as measured by Slow Vital Capacity (SVC).
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Verdiperstat | Matching Placebo
Number analyzed (Participants) | 126 | 122
percent change | -7.76 (1.519) | -8.05 (1.418)
Statistical Analysis 1: Comparison: Verdiperstat vs Matching Placebo; Test type: Superiority; p = 0.8875, Mixed Models Analysis; Covariates include baseline use of edaravone and riluzole, months since symptom onset, and pre-baseline ALSFRS-R slope; Mean Difference (Net) = 0.29, 95% CI 2-sided [-3.74 to 4.32], Standard Error of Mean 2.054 — Verdiperstat 24-week change from baseline relative to placebo 24-week change from baseline

4. Secondary Outcome: Muscle Strength
Description: Change in muscle strength over time as measured isometrically using hand-held dynamometry (HHD).
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Verdiperstat | Matching Placebo
Number analyzed (Participants) | 126 | 122
percent change | -23.24 (2.863) | -26.81 (2.682)
Statistical Analysis 1: Comparison: Verdiperstat vs Matching Placebo; Test type: Superiority; p = 0.3538, Mixed Models Analysis; Covariates include baseline use of edaravone and riluzole, months since symptom onset, and pre-baseline ALSFRS-R slope; Mean Difference (Net) = 3.57, 95% CI 2-sided [-3.99 to 11.13], Standard Error of Mean 3.848 — Verdiperstat 24-week change from baseline relative to placebo 24-week change from baseline

5. Secondary Outcome: Number of Participants That Experienced Death or Death Equivalent
Description: The number of participants who died or met the criterion for a death equivalent from the date of their baseline visit to the end of the Week 24 visit window (generally 175 days after baseline). The death equivalent criterion is use of permanent assisted ventilation (PAV) for more than 22 hours per day for more than 7 days in a row.
Time Frame: 24 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Verdiperstat | Matching Placebo
Number analyzed (Participants) | 126 | 122
Participants | 7 | 5
Statistical Analysis 1: Comparison: Verdiperstat vs Matching Placebo; Test type: Superiority; p = 0.318, Log Rank

ADVERSE EVENTS:
Time Frame: Up to 35 weeks after participant signed Master Protocol consent.
Arm/Group | Verdiperstat | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 6/126 | 0/41
Serious Adverse Events (participants affected / at risk) | 20/126 | 2/41
Other Adverse Events (participants affected / at risk) | 114/126 | 37/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verdiperstat (N=126) | Matching Placebo (N=41)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 2 (2) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Sudden death (General disorders) | 1 | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hepatic enzyme abnormal (Investigations) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verdiperstat (N=126) | Matching Placebo (N=41)
Headache (Nervous system disorders) | 27 (31) | 9 (11)
Muscular weakness (Nervous system disorders) | 22 (35) | 12 (18)
Neuromyopathy (Nervous system disorders) | 16 (22) | 8 (9)
Tension headache (Nervous system disorders) | 13 (17) | 3 (7)
Dizziness (Nervous system disorders) | 13 (15) | 3 (3)
Dysarthria (Nervous system disorders) | 4 (4) | 3 (4)
Nausea (Gastrointestinal disorders) | 35 (40) | 3 (3)
Constipation (Gastrointestinal disorders) | 24 (26) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 12 (13) | 4 (6)
Salivary hypersecretion (Gastrointestinal disorders) | 10 (10) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 10 (12) | 1 (1)
Fatigue (General disorders) | 20 (21) | 11 (14)
Oedema peripheral (General disorders) | 7 (8) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 24 (50) | 9 (16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1)
Insomnia (Psychiatric disorders) | 25 (28) | 0 (0)
Anxiety (Psychiatric disorders) | 9 (9) | 1 (1)
Urinary tract infection (Infections and infestations) | 10 (11) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 2 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (11) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4)
Blood thyroid stimulating hormone increased (Investigations) | 11 (12) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 8 (8) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 13 (13) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT04436510/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT04436510/SAP_001.pdf